CLINICAL TRIAL: NCT01522625
Title: Efficacy of Tenofovir Disoproxil Fumarate in Chronic Hepatitis B Patients With High Viral Load But Slight Aminotransferase Elevation
Brief Title: Tenofovir in Chronic Hepatitis B With Mild ALT Elevation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: E-DA Hospital (Other)
Collaborators: Gilead Sciences (Industry); Taipei Institute of Pathology (Other Government)
Responsible Party: Principal Investigator, Tu, Yuan-Kun, superintendent, E-DA Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMRP36100N
Record Dates: First submitted 2012-01-27; First posted 2012-01-31 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B; hepatitis B viral DNA; antiviral therapy; Tenofovir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- TDF (Experimental): tenofovir disoproxil fumarate (TDF) 300mg
  Interventions: Drug: tenofovir disoproxil fumarate 300mg per day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tenofovir disoproxil fumarate 300mg per day — tenofovir disoproxil fumarate 300mg per day for 3 years
  Other Names: Viread® (Gilead Sciences Inc)
  Arms: TDF
Drug: Placebo — Placebo, identical to TDF in appearance, once daily for 3years
  Arms: Placebo

SUMMARY:
This study aims to clarify whether patients with chronic hepatitis B with high viral load will benefit from oral antiviral therapy despite only mildly elevated serum liver enzyme.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) is a serious disease in Taiwan, leading to substantial morbidity and mortality including hepatic failure, liver cirrhosis, and hepatocellular carcinoma (HCC). Recently a large body of evidence supports that high level of serum HBV DNA is an independent risk factor for late complications in CHB patients. Nucleos(t)ide analogues (NUC) are effective antiviral therapy that can potently inhibit replication of hepatitis B virus (HBV), and has been widely used in management of patients with CHB. Current practice guidelines recommend using serum alanine aminotransferase (ALT) > 2 times of the upper limit of normal (ULN) as the prerequisite to initiate antiviral therapy in compensated CHB patients without liver cirrhosis. However, serum ALT level does not exactly correlate with serum HBV DNA or liver tissue injury. Whether antiviral therapy improves outcomes of patients with slightly elevated ALT (i.e. 1-2 folds of ULN) remains unknown.

ELIGIBILITY:
Inclusion Criteria:

* age between 25 to 70 years,
* serum HBsAg positivity for more than 6 months,
* positive or negative serum HBeAg,
* serum HBV DNA more than 2,000 IU/mL,
* highest serum ALT > 1 fold of ULN, but < 2 X ULN on at least two occasions (≧ 3 months apart) in the preceding one year,

Exclusion Criteria:

* co-infection with HIV, HCV, or HDV,
* previous exposure to HBV antiviral therapy for more than 12 weeks,
* presence of cirrhosis on histopathology,
* hepatic decompensation defined as serum bilirubin > 2mg/dl and prolonged prothrombin time > 3 seconds,
* concurrent malignant diseases including hepatocellular carcinoma,
* severe co-morbidity with life expectancy < 1year,
* pregnant or lactating women,
* organ transplantation except cornea or hair transplant,
* suspected or confirmed chronic liver diseases from etiologies other than HBV (e.g. alcoholic hepatitis, Wilson disease, Hemochromatosis…etc),
* serum creatinine >1.5mg/dL

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-01; Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Severity of hepatic necroinflammation and fibrosis | Within one month after completion of antiviral therapy
  Primary outcome is the severity of necroinflammation and fibrosis in liver tissue as evaluated by Knodell and Ishak scoring system

SECONDARY OUTCOMES:
Undetectable hepatitis B viral DNA | Within one month after completion of antiviral therapy
  HBV DNA viral DNA not detected in serum
Normalization of serum alanine aminotransferase | Within one month after completion of antiviral therapy
  serum ALT <40 IU/mL
Serum level of HBsAg | Within one month after completion of antiviral therapy
  quantification of serum HBV serface antigen
Serious adverse reaction | Within one month after completion of antiviral therapy
  Defined as death, life threatening event, permanent or temporary disability, and hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Chun Hsu, MD, MSc, Principal Investigator — E-Da Hospital, Kaohsiung, Taiwan; Jaw-Town Lin, MD, PhD, Study Chair — National Taiwan University
Locations (6):
- Taiwan (6):
  - Chia-Yi Christine Hospital, Chiayi City
  - E-Da Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Liouying, Tainan
  - Mackay Memorial Hosp, Taipei
  - National Taiwan University Hospital Yun-Lin Branch, Yunlin

REFERENCES:
- [Derived] Hsu YC, Chen CY, Chang IW, Chang CY, Wu CY, Lee TY, Wu MS, Bair MJ, Chen JJ, Chen CC, Tseng CH, Tai CM, Huang YT, Ku WH, Mo LR, Lin JT. Once-daily tenofovir disoproxil fumarate in treatment-naive Taiwanese patients with chronic hepatitis B and minimally raised alanine aminotransferase (TORCH-B): a multicentre, double-blind, placebo-controlled, parallel-group, randomised trial. Lancet Infect Dis. 2021 Jun;21(6):823-833. doi: 10.1016/S1473-3099(20)30692-7. Epub 2021 Jan 29. PMID 33524314